CLINICAL TRIAL: NCT04420390
Title: Low Dose Radiotherapy as Antinflammatory Treatment for COVID-19 Pneumonitis
Brief Title: Low Dose Radiotherapy for COVID-19 Pneumonitis
Acronym: LOWRAD-Cov19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital San Carlos, Madrid (Other)
Responsible Party: Principal Investigator, Manuel Gonzalo Vázquez Masedo, MD, PhD, Hospital San Carlos, Madrid
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LOWRAD-Cov19
Record Dates: First submitted 2020-05-14; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Covid19
Keywords: Radiotherapy; Antiinflammatory; Pneumonitis
MeSH Terms: conditions — COVID-19; Pneumonia | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiotherapy (Experimental)
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — Low-dose radiotherapy

SUMMARY:
SARS-CoV-2 is causing an unprecedented stress on healthcare systems around the world, due to its high rate of infection and the high morbidity and mortality.

The COVID-19 infection triggers an inflammatory cascade with cytokine synthesis, prompting the immune response. Low dose radiotherapy (LD-RT) (≤ 100 cGy) induces an anti-inflammatory response, lowering levels of pro-inflammatory cytokines such as IL-1β or inhibit leukocyte recruitment. LD-RT has been used historically for the pneumonia treatment reporting a rapid clinical improvement (within the first week), as well as a reduced mortality (from around 30% to 10%). Considering these results, LD-RT can potentially afford a therapeutic benefit against SARS-CoV-2. The study purpose is to evaluate prospectively the safety and efficacy of LD-RT for SARS-CoV-2.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 60 years.
2. COVID19 + confirmed by PCR.
3. Thoracic imaging study (chest X-ray, chest CT or PET-CT), compatible with lung involvement.
4. Phase II or lung phase without any improvement with pharmacological treatment.
5. Phase III or hyper-inflammatory phase without any improvement with pharmacological treatment
6. Poor clinical and functional respiratory evolution: > 30 breaths / minute, SpO2 <93%, PaO2 / FiO2 <300.
7. D-dimer> 1000 ng / mL or rising, ferritin> 1000 ng / mL, PCR> 10 mg / dL or double than before.

Exclusion Criteria:

1. Severe comorbidities that could hamper the radiation treatment.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-09-08 (Estimated)

PRIMARY OUTCOMES:
Radiological response | 3 days after low dose radiation
  Radiological results: Radiological worsening, improvement or without significant changes
Radiological response | 7 days after low dose radiation
  Radiological results: Radiological worsening, improvement or without significant changes

SECONDARY OUTCOMES:
Remission of respiratory symptoms | up to 6 months
  Remission of respiratory symptoms
SPO2 and PaO2/FiO2 | 7 days
  Time to SPO2>94% or PaO2/FiO2 >350mmHg without oxygen
Adverse events | 1 year
  Occurrence and grade of CTCAE 5.0 adverse events
Hospitalization | 3 months
  Duration of hospitalization
Overall survival | 1 month
  Overall survival
Ferritin value | 1 day after low dose radiation
  ferritin value (ng/mL)
Ferritin value | 2 days after low dose radiation
  ferritin value (ng/mL)
Ferritin value | 3 days after low dose radiation
  ferritin value (ng/mL)
blood cell count | 1 day after low dose radiation
  blood cell count (unit/L)
blood cell count | 2 days after low dose radiation
  blood cell count (unit/L)
blood cell count | 3 days after low dose radiation
  blood cell count (unit/L)
C-reactive protein | 1 day after low dose radiation
  C-reactive protein (mg/dl)
C-reactive protein | 2 days after low dose radiation
  C-reactive protein (mg/dl)
C-reactive protein | 3 days after low dose radiation
  C-reactive protein (mg/dl)
D-dimer | 1 day after low dose radiation
  D-dimer (ng/ml)
D-dimer | 2 days after low dose radiation
  D-dimer (ng/ml)
D-dimer | 3 days after low dose radiation
  D-dimer (ng/ml)
LDH levels | 1 day after low dose radiation
  LDH levels (UI/L)
LDH levels | 2 days after low dose radiation
  LDH levels (UI/L)
LDH levels | 3 days after low dose radiation
  LDH levels (UI/L)

CONTACTS AND LOCATIONS:
Locations (1):
- Servicio de Oncología Radioterápica. Hospital Clínico San Carlos, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No